CLINICAL TRIAL: NCT02577276
Title: Joint Gertner ReAbility Online and Mayo Clinic Feasibility Study: Evaluation of a Tele-Rehabilitation Service Program
Brief Title: Evaluation of a Tele-Rehabilitation Service Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: The Gertner Institute (Other); ReAbility Online (Other)
Responsible Party: Principal Investigator, Allen Brown, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-006308
Record Dates: First submitted 2015-10-12; First posted 2015-10-16 (Estimated); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Stroke; Paresis
Keywords: stroke; remote monitoring; hemiparesis
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tele-motion rehabilitation system (Experimental): Clinicians remotely monitor subjects' motor performance using Microsoft Kinect 3D sensor tracking system in their home to record their upper limb and trunk movements as they participate in a variety of functional tasks and motor activities, which are directed by their interaction with a monitor screen in their home using uniquely adapted software to integrate key rehabilitation intervention principles.
  Interventions: Device: Tele-motion rehabilitation system

INTERVENTIONS:
Device: Tele-motion rehabilitation system — Tele-motion rehabilitation system: Interventions include functional therapeutic exercise and real-time feedback. Clinicians remotely monitor subjects' motor performance using Microsoft Kinect 3D sensor tracking system in their home to record their upper limb and trunk movements as they participate in a variety of functional tasks and motor activities, which are directed by their interaction with a monitor screen in their home using uniquely adapted software to integrate key rehabilitation intervention principles.
  Other Names: Microsoft XB1 Kinect Sensor

SUMMARY:
Is a unique tele-rehabilitation service directed at treating upper limb weakness due to stroke feasible to provide at Mayo Clinic and are the individuals with stroke and the clinicians providing the care satisfied with the process?

DETAILED DESCRIPTION:
Participants will be identified from Mayo Clinic Division of Brain Rehabilitation's existing clinical practice and recruited either in person or by using a phone script.

Eligible participants will have 2 in-person clinical assessments, one before the intervention and one concluding the protocol. The first clinical assessment will involve introducing and familiarizing the participant with the study procedure, demonstrating and practicing with the system, and obtaining baseline clinical measures. During this first session the participant's technical skills and home equipment capabilities will be assessed and any assistance needed for establishing the technology in their home will be determined and provided. The second clinical assessment will include acquiring post-intervention clinical and outcome measures. Intervention duration will be 3 months. During the study period, each participant will receive online treatment for up to 45 minutes (in order to have net 30 min clinical time) twice per week. During these sessions, the clinician will teach system interaction including integrating feedback, instruct in system intervention activities and assure participant competence in system use, and adjust the level of difficulty in each activity according to the participant's abilities and needs. After the first month of intervention, the participant may be given permission by the therapist to train with the system for no more than 40 minutes per day. Such self-training opportunities are in addition to the twice weekly online sessions with the therapist.

ELIGIBILITY:
Inclusion

* >12 months after stroke
* Age 21-80 years
* A minimum of 45 degrees of flexion in the affected shoulder
* Active extension of the affected elbow to 150 degrees
* Independent sitting balance
* Able to understand simple instructions
* Lives within a 100 mile radius and able to attend two clinical assessments at Mayo Clinic
* Able to install the tele-rehabilitation software with minimal remote technical support
* Available caregiver as needed who has basic technical understanding of computer operation
* i3 processor based PC; 26" monitor; Windows 7 or 8 operating system; Internet connection of at least 10Mbps.

Exclusion

* Medical conditions that may limit physical activity at the level of low intensity cardio-vascular exercise
* Any contraindication related to the integrity of the musculoskeletal system
* Active malignancy
* Uncontrolled epilepsy
* Global aphasia
* Severe apraxia
* Severe ataxia
* Unilateral spatial neglect
* Chronic pain
* Pregnancy
* Adults lacking capacity

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-11-06 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Satisfaction Questionnaire | 3 months
  Clinician and participant satisfaction questionnaire
System Usability Scale | 3 months
  Clinician and participant usability questionnaire
Qualitative measure of technology/communications problems | 3 months
  Self report text of problems and difficulty with experimental technology and communication from participants and clinicians

SECONDARY OUTCOMES:
Upper limb (shoulder, elbow) range of motion | Baseline and at 3 months
  Upper limb (shoulder, elbow) range of motion of the participant as measured by a goniometer
Fugl- Meyer Scale | Baseline and at 3 months
  Fugl- Meyer Assessment for the participant's upper limb
Motor Activity Log (MAL) | Baseline and at 3 months
  Individuals are asked to rate Quality of Movement (QOM) and Amount of Movement (AOM) during 30 daily functional tasks (original MAL), 28 functional tasks (MAL 28) or 14 tasks (MAL 14). Target tasks include object manipulation (e.g. pen, fork, comb, and cup) as well as the use of the arm during gross motor activities (e.g. transferring to a car, steadying oneself during standing, pulling a chair into a table while sitting). Items scored on a 6-point ordinal scale.
Measures from the ReAbility Online system of participant and clinician activity | Weekly through 3-month study period
  Time of practice by participant as measured by the ReAbility Online system
Task performance scores | Weekly through 3-month study period
  Participant task performance scores as measured by the ReAbility Online system
Upper limb range of motion | Weekly through 3-month study period
  Upper limb range of motion of participant as measured by the ReAbility Online system
Number of compensatory movements | Weekly through 3-month study period
  Number of compensatory movements as measured by the ReAbility Online system
Time online | Weekly through 3-month study period
  Time online of participant and clinician as measured by the ReAbility Online system

CONTACTS AND LOCATIONS:
Overall Officials: Allen Brown, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No